CLINICAL TRIAL: NCT00869635
Title: Photodynamic Therapy With S-1 in the Patients With Unresectable Type III or IV Cholangiocarcinoma: A Prospective Randomized Trial With Open Label Control
Brief Title: S-1 and Photodynamic Therapy in Cholangiocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Do Hyun Park, Assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-0056
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Photodynamic therapy; S-1
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Treatment by combination of photodynamic therapy and S-1
  1. PDT with Photofrin® 2mg/kg i.v. 48hrs before laser activation
  2. S-1 chemotherapy before intolerable complication or definite tumor progression Based on the body surface area, <1.25m2: 80mg/day, 1.25~1.5m2: 100mg/day, ≧1.5m2: 120mg/day Given orally twice daily for 14days, followed by 7 days without treatment
  Interventions: Drug: S-1 Chemotherapy; Procedure: Photodynamic therapy
- 2 (Active Comparator): Treatment by photodynamic therapy only
  1. PDT with Photofrin® 2mg/kg i.v. 48hrs before laser activation
  2. Other managements except systemic chemotherapy were added freely.
  Interventions: Procedure: Photodynamic therapy
- 3 (Other): Treatment by photodynamic therapy only or combined chemotherapy with photodynamic therapy: Open label
  Interventions: Procedure: Photodynamic therapy; Procedure: Systemic chemotherapy except S-1

INTERVENTIONS:
Drug: S-1 Chemotherapy — S-1 chemotherapy before intolerable complication or definite tumor progression Based on the body surface area, <1.25m2: 80mg/day, 1.25~1.5m2: 100mg/day, ≧1.5m2: 120mg/day Given orally twice daily for 14days, followed by 7 days without treatment
  Arms: 1
Procedure: Photodynamic therapy — PDT with Photofrin® 2mg/kg i.v. 48hrs before laser activation
Procedure: Systemic chemotherapy except S-1 — Variable systemic chemotherapy except S-1
  Arms: 3

SUMMARY:
In patients with unresectable perihilar cholangiocarcinoma, photodynamic therapy with biliary stent has been known for palliation of jaundice and improving survival. But most of therapeutic effects were expected to delay bile duct obstruction rather than to decrease the tumor. Recently orally available chemotherapeutic agent, S-1 was reported as effective in patients with bile duct adenocarcinoma. The investigators' aims of study evaluate the combined effect of photodynamic therapy and S-1.

DETAILED DESCRIPTION:
In patients with unresectable perihilar cholangiocarcinoma, photodynamic therapy with biliary stent has been known for palliation of jaundice and improving survival. But most of therapeutic effects were expected to delay bile duct obstruction rather than to decrease the tumor. Recently orally available chemotherapeutic agent, S-1 was reported as effective in patients with bile duct adenocarcinoma. The investigators' aims of study evaluate the combined effect of photodynamic therapy and S-1.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of cholangiocarcinoma
* Not eligible for curative surgery
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or better
* No serious or uncontrolled concomitant medical illness
* Adequate bone marrow function (absolute neutrophil count ≧1,500 ul, platelet count ≧75,000/ul)
* Consent this study in letter

Exclusion Criteria:

* Another neoplasia
* Porphyria
* Pregnant or breastfeeding women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Compare overall survival time in patients with unresectable perihilar cholangiocarcinoma treated with photodynamic therapy combined with or without S-1 | 12 months after study start

SECONDARY OUTCOMES:
Compare the frequency of repeat photodynamic therapy | 6 months after study start
Compare the frequency of biliary tract decompressive interventions | 6 months after study start
Compare the frequency of hospitalization | 6 months after study start

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Park DH, Lee SS, Park SE, Lee JL, Choi JH, Choi HJ, Jang JW, Kim HJ, Eum JB, Seo DW, Lee SK, Kim MH, Lee JB. Randomised phase II trial of photodynamic therapy plus oral fluoropyrimidine, S-1, versus photodynamic therapy alone for unresectable hilar cholangiocarcinoma. Eur J Cancer. 2014 May;50(7):1259-68. doi: 10.1016/j.ejca.2014.01.008. Epub 2014 Jan 30. PMID 24485665